CLINICAL TRIAL: NCT05262374
Title: A Single Blinded Randomised Controlled Trial Comparing the Ergonomics of Laparoscopic and Versius Robotic Assisted Inguinal Hernia Surgery
Brief Title: Versius or Laparoscopic TransAbdominal Inguinal Hernia REpair
Acronym: VOLTAIRE
Status: Completed | Type: Observational
Sponsor: Milton Keynes University Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: MKUH-RD-021
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Inguinal Hernia
Keywords: surgery; ergonomics; robotics
MeSH Terms: conditions — Hernia, Inguinal | interventions — Laparoscopy; Robotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Laparoscopic Arm: This cohort of participants will have their procedure completed by a human surgeon
  Interventions: Procedure: Procedure/Surgery: Laparoscopic
- Robotic Arm: This cohort of participants will have their procedure completed by the Versius Surgical Robotic System.
  Interventions: Procedure: Robotic

INTERVENTIONS:
Procedure: Procedure/Surgery: Laparoscopic — Surgeon
  Groups: Laparoscopic Arm
Procedure: Robotic — Versius system.
  Groups: Robotic Arm

SUMMARY:
This trial will compare laparoscopic and robotic-assisted inguinal hernia repairs, using the Versius® system. We will initially aim to recruit 60 patients (20 patients in the laparoscopic arm and 40 in the robotic arm) in order to assess the ergonomic impact of each modality on the operating surgeon. This aims to provide in vivo information on whether robotic surgery provides any advantages to the operating surgeon. This trial will also be used to assess the feasibility of recruitment to a future larger study, and any data collected will be used as pilot data.

DETAILED DESCRIPTION:
This study has been designed to assess the ergonomics of Versius® assisted surgery in comparison with laparoscopic surgery in the management of inguinal hernias. The study will randomise 60 patients who require repair of an inguinal hernia and have been deemed suitable for a minimally invasive approach. Patients will be randomised to receive either laparoscopic or Versius® robotic assisted surgery but will be informed that it will be attempted via a minimally invasive approach that could include either of these two subtypes of minimally invasive surgery. The randomisation will occur on a 2:1 basis, with 2 patients allocated to the robotic arm for every 1 patient allocated to the laparoscopic arm. Laparoscopic surgery is already a well-established technique, and therefore the study team believe more valuable data about the outcomes of robotic surgery will be obtained with this randomisation ratio given that no prior studies have been undertaken using this robotic platform. All surgeons in the study will be required to have been involved in at least 20 cases performed using the relevant modality, whether for the robotic or laparoscopic cohorts.

Data will be collected at four key timepoints; recruitment, intraoperatively, at discharge and again at 14 days following intervention. Feasibility outcomes will include willingness to be recruited to study (acceptability), willingness for patient to undergo desired randomised operative approach (acceptability/concordance), withdrawal of patients (non-concordance), study retention (retention rates), and the usefulness and limitations of outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Need for inguinal hernia repair surgery
* Deemed suitable for minimally invasive surgery

Exclusion Criteria:

* Patients who are unable to consent
* Prisoners
* Patients in need of emergency surgery
* Patients with inguinoscrotal or recurrent inguinal hernias

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who require surgery to repair an inguinal hernia will be approached to participate in the trial.
  In this trial, all patients will be only be considered if deemed suitable for surgery via a minimally invasive approach
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
To compare the operating surgeon ergonomics (physical strain) of laparoscopic and Versius® robotic assisted surgery | Length of the procedure expected to be between 1-4 hours
  body position (physical strain) and cognitive workload (mental strain) assessed using the REBA score

SECONDARY OUTCOMES:
Measurement of the rate of participant recruitment | Through study completion, an average of 1 year.
  Measure the number of participants recruited over the length of time. The units of measurement will be presented on a scale of number of participants over a predetermined length of time
Measurement of drop-out (withdrawal) rate of participants | Assessed from Day 1 (Randomisation) to date of withdrawal
  Measure the number of participants who withdrawal (drop out) from the trial. The units of measurement will be presented on a scale of numbers of withdrawals versus time.
Measurement of the unblinding rate of participants | Through study completion, an average of 1 year.
  Measure the number of participants where the treatment is unblinded during the trial. This is measured by the number of participants over the length of time who's treatment is unblinded.
Mental strain of surgeon | 30 minutes maximum completion time per surgeon
  To compare the operating surgeon mental strain of each approach using the NASA-Task Load Index score.
Health Economics | Procedure and recovery inpatient stay per participant expected to be between 1-3 days.
  Explore health economic aspects of each approach via calculation of the entire hospital episode and individual operation (including fixed costs and instrument costs) comparing the cost for cohort using the Versus Surgical Robot versus the human surgeon.
Communication | 1-4 hours expected for the duration of the procedure
  To compare differences in in-theatre communication assessed from audiovisual footage, using the Oxford NOTECHS II score.
Satisfaction with life scale | Assessed on Day 1 and Day 14
  Quality of life units completion of EQ-5D-5L questionnaires post operatively at recruitment Day 1 and on day 14. Total scores used not sub scales to be reported.
Satisfaction with life | Assessed on Day 1 and Day 14
  Quality of life units completion of MFSI-SF questionnaires post operatively at recruitment Day 1 and on day 14. Total scores used not sub scales to be reported.
Length of in-patient stay | Through study completion, an average of 1 year
  Measure of the time in days of each participant's hospital stay as an in-patient.
Pain Scores | Day 14
  Using a uni-dimensional pain score measurement examining the change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Barrie Keeler, Principal Investigator — Colorectal surgeon
Locations (1):
- Surgical Division, Milton Keynes, United Kingdom

IPD SHARING:
Plan to Share IPD: No